CLINICAL TRIAL: NCT05774717
Title: Tranexamic Acid in Rhinoplasty: Perioperative Bleeding, Edema and Ecchymosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Shiayin Yang, Assistant Professor of Otolaryngology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 221035
Record Dates: First submitted 2022-10-12; First posted 2023-03-20 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Surgery; Postoperative Blood Loss
MeSH Terms: conditions — Postoperative Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: One group receives tranexamic acid prior to surgery, one group receives nothing (routine care).
Masking Description: Provider will order tranexamic acid based based on even versus odd last digit of medical record number (MRN). Patient will be blinded, as will all personnel analyzing postoperative photographs and other data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tranexamic Acid (Experimental): Patients receive 1 gram IV tranexamic acid in the operating room prior to surgical incision.
  Interventions: Drug: Tranexamic acid
- Control (No Intervention): Routine care, no tranexamic acid given.

INTERVENTIONS:
Drug: Tranexamic acid — 1 gram IV (intravenous) tranexamic acid administered in the operating room just prior to starting the case (10 minutes), at time that routine preoperative antibiotic is given.
  Other Names: TXA
  Arms: Tranexamic Acid

SUMMARY:
This study will be a prospective randomized study to evaluate the effect of tranexamic acid (TXA) use on intraoperative and postoperative outcomes among patients undergoing rhinoplasty by two Facial Plastic surgeons at Vanderbilt. Outcomes will include intra- and post-operative bleeding and postoperative bruising and swelling.

DETAILED DESCRIPTION:
TXA is an antifibrinolytic agent that acts to decrease bleeding by stabilizing the fibrin matrix involved in the clotting cascade. The use of TXA, oral or intravenous, has been extensively used and described in the literature to prevent exsanguination in trauma and in various surgical procedures, as well as for heavy menstrual bleeding. It has been used in the perioperative period during various nasal and sinus surgery, and current research in rhinoplasty suggests that its use may decrease intraoperative bleeding and postoperative eye swelling and bruising.

Currently, IV TXA is used at this institution in some cases by some surgeons in the perioperative period in rhinoplasty surgery, though its used is not standardized and has not been studied. This study will randomize patients undergoing rhinoplasty, with consent, to receive TXA or placebo in the perioperative period. The investigators anticipate collecting 60-100 patients. Outcomes will include intraoperative bleeding, postoperative swelling and bruising (both subjective and based on blinded reviewer analysis of postoperative photographs).

TXA has been used in the perioperative period during various nasal and sinus surgery, and current research in rhinoplasty suggests that its use may decrease intraoperative bleeding and postoperative eye swelling and bruising. In these studies, TXA has been given in intravenous and/or oral form in 1-3 doses in the perioperative period, and there have been no serious adverse effects reported. IV TXA is also FDA approved for use at time of tooth extraction to decrease bleeding, and PO TXA is approved use during the menstrual cycle to decrease heavy menstrual bleeding. There are countless studies in the literature supporting use of both IV and PO TXA in trauma, orthopedic and spine surgery and neurosurgery, and it is widely used in clinical practice in these disciplines. It's use in rhinoplasty is growing, yet has not been studied in larger groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years of age who elect to undergo cosmetic or functional open primary rhinoplasty with osteotomies (repositioning the nasal bones) by Drs. Yang or Patel at VUMC.
* No other facial plastics procedure nor sinus surgery performed simultaneously
* Lack all the below Exclusion Criteria

Exclusion Criteria:

* Known allergy to TXA (tranexamic acid)
* Intracranial bleeding
* Known defective color vision
* History of venous or arterial thromboembolism
* Active thromboembolic disease
* Severe renal impairment (diagnosis of chronic kidney disease)
* History of coagulation disorder
* Known thrombocytopenia (platelets <150,000)
* Current use of anticoagulant (blood thinner)
* Uncontrolled DM (diabetes mellitus) preventing use of dexamethasone in the perioperative period
* Cardiac arrhythmia
* History of AMI (acute myocardial infarction), stroke, seizure, liver failure
* Laboratory results showing platelets <150,000, PT (prothrombin time) >45, INR (international normalized ratio) >1.2, seizure disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative bleeding as measured by the weight of surgical sponges used | During surgery
  Weight of surgical sponges used (grams)
Intraoperative bleeding as measured by the volume of blood in suction canister | Intraoperative
  Volume of blood in suction canister (Milliliters)
Postoperative bleeding as measured by patient-rated bleeding on Visual Analog Scale (VAS) | Up to one week following surgery.
  A single patient-answered question visual analog scale (VAS) used to measure the amount of post-operative bleeding from the nose the participant experienced (1 to 5 scale with 5 being the most)
Postoperative edema | Up to one week following surgery
  Swelling around the eyes (Visual Analog Scale, 1 to 5 scale with 5 being the most)
Postoperative ecchymosis | Up to one week following surgery
  Bruising around the eyes (Visual Analog Scale, 1 to 5 scale with 5 being the most)
Postoperative bleeding as measured by the number of medical interventions needed to control bleeding | Up to one week following surgery
  Number of interventions required to control bleeding (surgical or procedural interventions)

CONTACTS AND LOCATIONS:
Overall Officials: Shiayin F Yang, MD, Principal Investigator — Vanderbilt University Medical Center; Jaclyn S Lee, MD, Study Director — Vanderbilt University Medical Center; Alexander J Barna, MPH, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
No plan at this time to share.

REFERENCES:
- [Background] Avci H. The Effect of Different Dose Regimens of Tranexamic Acid in Reducing Blood Loss in Rhinoplasty: A Prospective Randomized Controlled Study. J Craniofac Surg. 2021 Jul-Aug 01;32(5):e442-e444. doi: 10.1097/SCS.0000000000007247. PMID 33208696
- [Background] de Vasconcellos SJA, do Nascimento-Junior EM, de Aguiar Menezes MV, Tavares Mendes ML, de Souza Dantas R, Martins-Filho PRS. Preoperative Tranexamic Acid for Treatment of Bleeding, Edema, and Ecchymosis in Patients Undergoing Rhinoplasty: A Systematic Review and Meta-analysis. JAMA Otolaryngol Head Neck Surg. 2018 Sep 1;144(9):816-823. doi: 10.1001/jamaoto.2018.1381. PMID 30098161
- [Background] Zaman SU, Zakir I, Faraz Q, Akhtar S, Nawaz A, Adeel M. Effect of single-dose intravenous tranexamic acid on postoperative nasal bleed in septoplasty. Eur Ann Otorhinolaryngol Head Neck Dis. 2019 Nov;136(6):435-438. doi: 10.1016/j.anorl.2018.10.019. Epub 2019 Jun 14. PMID 31204198
- [Background] Locketz GD, Lozada KN, Bloom JD. Tranexamic Acid in Aesthetic Facial Plastic Surgery: A Systematic Review of Evidence, Applications, and Outcomes. Aesthet Surg J Open Forum. 2020 Jun 14;2(3):ojaa029. doi: 10.1093/asjof/ojaa029. eCollection 2020 Sep. PMID 33791652
- [Background] Jouybar R, Nemati M, Asmarian N. Comparison of the effects of remifentanil and dexmedetomidine on surgeon satisfaction with surgical field visualization and intraoperative bleeding during rhinoplasty. BMC Anesthesiol. 2022 Jan 14;22(1):24. doi: 10.1186/s12871-021-01546-9. PMID 35031005